CLINICAL TRIAL: NCT00690911
Title: A Phase II, Multi-Center, Open Label Study to Determine the Efficacy of Adalimumab in the Treatment of Cutaneous Sarcoidosis (HUM 04-36)
Brief Title: Study to Determine the Efficacy of Adalimumab in the Treatment of Cutaneous Sarcoidosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dr. Jorizzo has decided to withdraw from this study due to the time it is taking to get the study started.
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00002161; 32409
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): open label adalimumab 40mg
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — 40mg dose subcutaneously using sterile technique. The site research staff will instruct and supervise subjects or a designee or nurse on proper injection technique during site visit evaluations. Subjects or a reliable designee will administer injectable study drug at home in between site visit evaluations.
  Other Names: Humira

SUMMARY:
The purpose of the study is to see if Humira is effective and safe in the treatment of sarcoidosis.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and efficacy of adalimumab for the treatment of cutaneous sarcoidosis. A secondary objective is to study gene expression in sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject has a diagnosis of cutaneous sarcoidosis for greater than 6 months with a physician global assessment score of at least 4. Diagnosis (based on the recommendations of an expert panel 24) can be made by either:
* Skin lesions characteristic of sarcoidosis and a biopsy showing granulomas with no evidence of mycobacteria, fungus, or malignancy.
* A biopsy that does not show granulomas, but the patient has characteristic skin lesions and another clinical feature suggesting sarcoidosis (bilateral hilar adenopathy, erythema nodosum, uveitis, raised ACE level, BAL lymphocytosis (CD4:CD8>3.5), panda/lambda sign on gallium scan)
* If female of childbearing potential, subject will have a negative urine pregnancy test at Screening and Week 0.
* If female, subject will be either post-menopausal for > 1 year, surgically sterile (hysterectomy or bilateral tubal ligation), or practicing one form of birth control (abstinence, oral contraceptive, estrogen patch, implant contraception, injectable contraception, IUD, diaphragm, condom, sponge, spermicides, or vasectomy of partner). Female subjects will continue to use contraception for 6 months following the last infusion.
* Screening laboratory results are within the study parameters.
* Subject has been on a stable dose of antibiotics, thalidomide, antimalarials, oral corticosteroids or other immunosuppressives, such cyclosporine, tacrolimus, azathioprine, methotrexate, or mycophenolate mofetil over the previous 4 weeks.

Exclusion Criteria:

* Subject has evidence of a clinically significant, unstable or poorly controlled medical condition including unstable systemic sarcoidosis.
* Subject has a chest X-ray consistent with an active infection or previous exposure to TB and/or a positive purified protein derivative test at screening (>5 mm).
* Subject has a serious, active or recurrent bacterial, viral, or fungal infection. This includes hepatitis B and C, and HIV.
* Subject has been hospitalized for infection or received IV antibiotics within the previous 2 months prior to baseline.
* Subject has a history of tuberculosis at anytime or close contact with a person with active tuberculosis within the previous 6 months.
* Subject has received a live vaccination within the previous 3 months.
* Subject has a history of a central nervous system disorder/demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis.
* Subject has current signs or symptoms or history of systemic lupus erythematosus.
* Subject has been diagnosed with a malignancy within the past 5 years except for successfully treated non-melanoma skin cancer.
* Subject has signs or symptoms suggestive of a possible lymphoproliferative disease.
* Subject has a diagnosis of severe congestive heart failure (Class III or IV NYHA).
* Subject has had a substance abuse problem within the previous 3 years.
* Subject has any dermatologic disease in the target site that may be exacerbated by treatment or interfere with examination.
* Subject has been treated with an anti-TNF biologic immune response modifier, such as infliximab, adalimumab, or etanercept within the past 8 weeks.
* Subject has been treated with topical corticosteroids, tacrolimus, or pimecrolimus within 2 weeks or intralesional corticosteroids within 4 weeks of baseline.
* Subject has been administered an investigational drug in another clinical study within 30 days prior to baseline (or 5 half-lives, whichever is longer).
* Subject has a known allergy to adalimumab.
* Subject is female and is pregnant, is considering becoming pregnant during the study and for 6 months afterwards, or is nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in PGA score. | 24 weeks

SECONDARY OUTCOMES:
Number of complete responders, partial responders, minimal responders, and non-responders | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jorizzo, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States